CLINICAL TRIAL: NCT04709484
Title: Comparison of the Effectiveness of USG and Palpation Guidance Steroid Injection in Patients With Plantar Fasciitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sultan Abdulhamid Han Training and Research Hospital, Istanbul, Turkey (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: dr.ademerbirol
Record Dates: First submitted 2021-01-12; First posted 2021-01-14 (Actual); Results first posted 2021-10-20 (Actual); Last update posted 2021-10-20 (Actual); Status verified 2021-10

CONDITIONS: Plantar Fasciitis
Keywords: Plantar Fasciitis; USG; Steroid; Injection
MeSH Terms: conditions — Fasciitis, Plantar

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: double(participant, outcomes assesor double)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- USG-guided steroid injection group (Experimental): In the USG-guided group, steroid injection will be made to the area where the fascia is thickened under USG guidance. The content of the steroid solution will be 1 ml of 1% Lidocaine + 1 ml (40 mg) methylprednisolone.
  Interventions: Drug: USG-guided steroid injection
- Palpation-guided steroid injection group (Experimental): In the palpation-guided group, the most painful point will be found by palpation on the calcaneus bone and steroid injection will be made to that part. The content of the steroid solution will be 1 ml of 1% Lidocaine + 1 ml (40 mg) methylprednisolone.
  Interventions: Drug: Palpation-guided steroid injection

INTERVENTIONS:
Drug: USG-guided steroid injection — In the palpation-guided group, the most painful point will be found by palpation on the calcaneus boIn the USG-guided group, steroid injection will be made to the area where the fascia is thickened under USG guidance. The content of the steroid solution will be 1 ml of 1% Lidocaine + 1 ml (40 mg) methylprednisolone.ne and steroid injection will be made to that part. The content of the steroid solution will be 1 ml of 1% Lidocaine + 1 ml (40 mg) methylprednisolone.
  Other Names: no other names
  Arms: USG-guided steroid injection group
Drug: Palpation-guided steroid injection — In the palpation-guided group, the most painful point will be found by palpation on the calcaneus bone and steroid injection will be made to that part. The content of the steroid solution will be 1 ml of 1% Lidocaine + 1 ml (40 mg) methylprednisolone.
  Other Names: no other names
  Arms: Palpation-guided steroid injection group

SUMMARY:
Plantar fasciitis, often described as overloading of the plantar fascia, is the most common cause of heel pain in adults. It is characterized by a sharp pain along the medial aspect of the heel, which is worse with the first step taken in the morning or at the beginning of an activity and decreases as the person warms up. The etiology of plantar fasciitis is multifactorial and not well understood. Poor biomechanics and changes in the structure of the foot can lead to repeated micro-trauma at the beginning of the plantar fascia, causing inflammation and degeneration. Plantar fasciitis is more common in sedentary individuals and athletes and those participating in running sports. Other risk factors associated with plantar fasciitis include reduced ankle dorsiflexion, increased body mass index (BMI), and work-related weight loss activities.

Current treatments for plantar fasciitis, such as plantar fascia stretching exercises, strapping, extracorporeal shock wave therapy, nonsteroidal anti-inflammatory drugs (NSAIDs), arch braces, and heel pads are mainly aimed at reducing inflammation. Corticosteroid injections are usually reserved for refractory plantar fasciitis after conservative noninvasive attempts have failed. It has been shown to effectively reduce heel pain in patients with plantar fasciitis. The strong anti-inflammatory effect of corticosteroids can speed up the process of pain relief.

In our study, we aimed to compare the effectiveness of USG and palpation guidance blind steroid injection in patients diagnosed with plantar fasciitis.

DETAILED DESCRIPTION:
It is planned to enroll 60 (sixty) patients in the study. Patients diagnosed with plantar fasciitis, between the ages of 18-75, who have failed conservative treatment (stretching exercises, non-steroidal anti-inflammatory drugs and heel pads) for at least 3 months, and those with a Visual Anolog Scale value of 5 and above will be included in the study. Any local injection therapy and physical therapy for heel pain in the last 4 months, any surgery history for heel pain, history of tarsal tunnel syndrome, ankle effusion showing intra-articular disease, healed calcaneal fracture, Achilles tendinopathy, foot including pes and any deformity of the ankle, planus or pes cavus deformity; Patients with systemic disorders such as diabetes mellitus, rheumatoid arthritis, hematological disease or gout, pregnancy, history of aspirin or aspirin-like medication, and mental insufficiency will be excluded from the study.

In the study, the patients will be filled in Visual Analogue Scale (VAS) and Foot Function Indez (FFI) questionnaires. Patients will be randomized into 2 groups according to the Random Number Generation. The first group will be the USG-guided steroid injection group, and the second group will be the palpation-guided steroid injection group. In the USG-guided group, steroid injection will be made to the area where the fascia is thickened under the guidance of USG. In the palpation-guided group, the most painful point will be found by palpation on the calcaneus bone and steroid injection will be made to that part. The content of the steroid solution will be 1 ml of 1% Lidocaine + 1 ml (40 mg) methylprednisolone. There will be pre-injection, 1st month and 3rd month controls after injection.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with plantar fasciitis
2. Between the ages of 18-75
3. Who have failed conservative treatment (stretching exercises, non-steroidal anti-inflammatory drugs and heel pads) for at least 3 months
4. Visual Anolog Scale value of 5 and above will be included in the study.

Exclusion Criteria:

1. Having received any local injection therapy and physical therapy for heel pain within the last 4 months,
2. Any history of surgery for heel pain, tarsal tunnel syndrome, calcaneal fracture, Achilles tendinopathy, any deformity of the foot and ankle including pes, planus or pes cavus deformity
3. with systemic disorders such as diabetes mellitus, rheumatoid arthritis, hematological disease, or gout
4. Pregnancy
5. A recent history of aspirin or aspirin-like medication
6. mental disability

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2021-03-11 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adem Erbirol, Study Director — Egirdir Bone Joint Diseases Treatment And Rehabilitation Hospital
Locations (1):
- Adem ERBİROL, Isparta, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
other researchers would get information from the main researcher. therefore it was not shared.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | USG-guided Steroid Injection Group | Palpation-guided Steroid Injection Group
Started | 34 | 32
Completed | 34 | 32
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | USG-guided Steroid Injection Group | Palpation-guided Steroid Injection Group | Total
Number analyzed (Participants) | 34 | 32 | 66
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 31 | 31 | 62
  >=65 years | 3 | 1 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.12 (8.29) | 48.78 (9.76) | 47.92 (9.00)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 29 | 58
  Male | 5 | 3 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 34 | 32 | 66
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Turkey | 34 | 32 | 66
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 29.92 (4.47) | 29.71 (4.81) | 29.82 (4.61)

OUTCOME MEASURES:

1. Primary Outcome: Pain Severity
Description: visual analog scale (0-10) minimum score: 0 maximum score: 10. Higher scores reflect more severe pain. Higher values represent a worse outcome.
Time Frame: day 0 (before intervention)
Population: intent to treat population(all participants)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | USG-guided Steroid Injection Group | Palpation-guided Steroid Injection Group
Number analyzed (Participants) | 34 | 32
score on a scale | 8.50 (0.90) | 8.31 (0.90)

2. Primary Outcome: Pain Severity
Description: as for outcome 1
Time Frame: 1 month after intervention
Population: intent to treat population(all participants)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | USG-guided Steroid Injection Group | Palpation-guided Steroid Injection Group
Number analyzed (Participants) | 34 | 32
score on a scale | 1.50 (1.83) | 1.53 (2.29)

3. Primary Outcome: Pain Severity
Description: as for outcome 1
Time Frame: 3 month after intervention
Population: intent to treat population(all participants)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | USG-guided Steroid Injection Group | Palpation-guided Steroid Injection Group
Number analyzed (Participants) | 34 | 32
score on a scale | 1.44 (2.08) | 1.75 (2.46)

4. Secondary Outcome: Foot Function Index
Description: Foot Function Index(FFI) is a self-report questionnaire concerning foot function and pain. The FFI consists of 23 questions with scores 0-10 in three domains concerning foot pain, function and disability resulting in a total score range from 0 to 230. The score is validated for patients with plantar fasciitis with a minimal clinical important difference being 7 points. Higher values represent a worse outcome.
Time Frame: day 0 (before intervention)
Population: intent to treat population(all participants)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | USG-guided Steroid Injection Group | Palpation-guided Steroid Injection Group
Number analyzed (Participants) | 34 | 32
score on a scale | 65.41 (12.78) | 63.78 (13.80)

5. Secondary Outcome: Foot Function Index
Description: as for outcome 4
Time Frame: 1 month after intervention
Population: intent to treat population(all participants)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | USG-guided Steroid Injection Group | Palpation-guided Steroid Injection Group
Number analyzed (Participants) | 34 | 32
score on a scale | 8.06 (13.46) | 7.47 (13.66)

6. Secondary Outcome: Foot Function Index
Description: as for outcome 4
Time Frame: 3 month after intervention
Population: intent to treat population(all participants)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | USG-guided Steroid Injection Group | Palpation-guided Steroid Injection Group
Number analyzed (Participants) | 34 | 32
score on a scale | 9.32 (14.15) | 8.41 (14.53)

ADVERSE EVENTS:
Time Frame: adverse events were not monitored/assessed
Description: adverse events were not monitored/assessed
Arm/Group | USG-guided Steroid Injection Group | Palpation-guided Steroid Injection Group
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-03-01): https://cdn.clinicaltrials.gov/large-docs/84/NCT04709484/Prot_000.pdf
  • Statistical Analysis Plan (2021-08-01): https://cdn.clinicaltrials.gov/large-docs/84/NCT04709484/SAP_001.pdf